CLINICAL TRIAL: NCT02624986
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Obinutuzumab in Combination With Idasanutlin in Patients With Relapsed or Refractory Follicular Lymphoma and Obinutuzumab or Rituximab in Combination With Idasanutlin in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Study of Idasanutlin in Combination With Obinutuzumab in Relapsed/Refractory (R/R) Follicular Lymphoma (FL) and in Combination With Rituximab in R/R Diffuse Large B-Cell Lymphoma (DLBCL) Participants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the study after Phase 1; will not proceed with Phase 2.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH29812; 2015-002100-83 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-04

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — RG7388; obinutuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 100 milligrams (mg) orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Obinutuzumab
- DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab
- DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 200 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab
- DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) in this bridging cohort received induction treatment with idasanutlin 150 mg orally in combination with rituximab 375 milligrams per square meter of body surface area (mg/m^2) IV for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Rituximab
- DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) in this bridging cohort received induction treatment with idasanutlin 200 mg orally in combination with rituximab 375 mg/m^2 IV for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Rituximab
- FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (Experimental): Participants with follicular lymphoma (FL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 100 milligrams (mg) orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab
- FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (Experimental): Participants with follicular lymphoma (FL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab
- FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (Experimental): Participants with follicular lymphoma (FL) in this bridging cohort received induction treatment with single-agent obinutuzumab 1000 mg IV for Cycle 1 and then idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for Cycles 2-6 (1 cycle = 28 days).
  Interventions: Drug: Idasanutlin; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Idasanutlin — Participants received idasanutlin film-coated tablets orally at a starting dose of 100 mg daily on Days 1 to 5 of each 28-day cycle. Escalation was to occur in at least 50-mg increments, and daily doses greater than or equal to (≥) 400 mg will be split into twice daily dosing.
  Other Names: RO5503781
  Arms: DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2; DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2; DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg; DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg; FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg; FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg; FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Drug: Obinutuzumab — Participants received a fixed dose of obinutuzumab 1000 mg intravenous (IV) infusion to be given on Days 1, 8 and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6 (1 cycle = 28 days). For eligible participants with FL, post-induction treatment was to be given at a dose of 1000 mg via IV infusion on Day 1 once every 2 months for a maximum of up to 24 months.
  Other Names: RO5072759
  Arms: DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg; DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg; DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg; FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg; FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg; FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Drug: Rituximab — Participants received a fixed dose of rituximab, 375 mg/m^2 IV infusion on Day 1 of Cycles 1-6. Post-induction treatment for eligible participants was to be given at a dose of 375 mg/m^2 IV infusion on Day 1 of every other month for up to 6 months, until disease progression or unacceptable toxicity.
  Other Names: RO0452294
  Arms: DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2; DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2

SUMMARY:
This is a open-label, multicenter, non-randomized, study to evaluate the safety, efficacy, and pharmacokinetics of idasanutlin in combination with obinutuzumab in participants with R/R FL and rituximab in combination with idasanutlin in R/R DLBCL. The study will include an initial dose-escalation phase followed by an expansion phase. The dose-escalation phase is designed to determine the recommended phase 2 dose (RP2D) for idasanutlin in combination with obinutuzumab for FL and in combination with rituximab for DLBCL. The expansion phase is designed to further assess the safety and efficacy of obinutuzumab in combination with idasanutlin at the RP2D with the selected regimen in participants with R/R FL and of rituximab in combination with idasanutlin at the RP2D in participants with R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Histologically documented cluster of differentiation (CD) 20-positive B-cell lymphoma classified as relapsed or refractory FL or DLBCL after treatment with at least two prior chemoimmunotherapy regimens that included an anti-CD20 monoclonal antibody (mAb) and for which no other more appropriate treatment option exists
* At least one bidimensionally measurable lesion
* Agreement to remain abstinent or use adequate contraception, among women or men of childbearing potential

Exclusion Criteria:

* Known CD20-negative status at relapse or progression
* Prior allogeneic stem cell transplantation (SCT), or autologous SCT within 100 days prior to Day 1 of Cycle 1
* Current use of systemic corticosteroids greater than (>) 20 mg prednisone per day (or equivalent), or prior anti-cancer therapy to include: radioimmunoconjugate within 12 weeks; mAb or antibody-drug conjugate within 4 weeks; or radiotherapy/chemotherapy/hormone therapy/targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1
* Requirement for chronic anticoagulation
* Central nervous system (CNS) disease
* Active infection
* Positive for human immunodeficiency virus (HIV) or hepatitis B or C
* Receipt of a live virus vaccine within 28 days prior to Day 1 of Cycle 1
* Poor hematologic, renal, or hepatic function
* Pregnant or lactating women
* History of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (8):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Colorado, Aurora, Colorado
  - Norton Medical Plaza II, Louisville, Kentucky
  - Swedish Cancer Institute, Cary, North Carolina
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Germany (5):
  - Zentralklinikum Augsburg, Augsburg
  - Charité Research Organisation GmbH Campus-Virchow-Klinikum, Berlin
  - Universitätsklinikum Köln, Cologne
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitätsklinikum Wurzburg, Würzburg
- New Zealand (3):
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Auckland Clinical Studies Limited, Grafton
- South Korea (5):
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 patients were screened, twenty-five of whom were enrolled in the dose escalation phase. The sponsor decided to terminate the study early and the expansion phase was not opened.
Groups:
- DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 100 milligrams (mg) orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
- DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
- DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 200 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
- DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) in this bridging cohort received induction treatment with idasanutlin 150 mg orally in combination with rituximab 375 milligrams per square meter of body surface area (mg/m^2) IV for 6 cycles (1 cycle = 28 days).
- DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) in this bridging cohort received induction treatment with idasanutlin 200 mg orally in combination with rituximab 375 mg/m^2 IV for 6 cycles (1 cycle = 28 days).
- FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory follicular lymphoma (FL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 100 milligrams (mg) orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
- FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory follicular lymphoma (FL) in this non-bridging dose-escalation cohort received induction treatment with idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
- FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory follicular lymphoma (FL) in this bridging cohort received induction treatment with single-agent obinutuzumab 1000 mg IV for Cycle 1 and then idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for Cycles 2-6 (1 cycle = 28 days).
Period: Overall Study
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Started (Intent-to-Treat (ITT) Population) | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Received Any Study Treatment (Safety Population) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Not completed — Death | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 1 | 1 | 0 | 1 | 2 | 2 | 4 | 3
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | Total
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (6.4) | 70.7 (15.2) | 55.5 (10.6) | 67.3 (8.4) | 56.5 (12.9) | 52.5 (6.4) | 53.3 (6.7) | 64.2 (9.8) | 60.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 4 | 12
  Male | 1 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 2 | 2 | 3 | 2 | 4 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 0 | 2 | 3 | 1 | 1 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response at the End of Induction, Determined by an Independent Review Committee (IRC) on the Basis of Positron Emission Tomography and Computed Tomography (PET-CT) Scans Using Modified Lugano 2014 Criteria
Description: The plan was for the IRC to evaluate responses at the end of induction treatment in participants from the expansion phase using Lugano 2014 criteria for malignant lymphoma for a PET-CT-based complete response (CR), which required a complete metabolic response with a score of 1, 2, or 3 with or without a residual mass in lymph nodes and extralymphatic sites on the PET 5-point scale for 18-fluorodeoxyglucose (FDG) uptake (1 = no uptake above background; 2 = uptake less than or equal to [≤] mediastinum; 3 = uptake greater than [>] mediastinum and ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly > liver and/or new lesions). The CR criteria were slightly modified to require normal bone marrow by morphology (if indeterminate, immunohistochemistry negative). PET-CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: The study plan was for the IRC to analyze the efficacy results in participants from the expansion phase (Phase 2), but the expansion phase was not opened (i.e., no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Phase 1).
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With a Dose-Limiting Toxicity
Description: A dose-limiting toxicity (DLT) was defined as at least one of the following events occurring during Cycle 1 (or first 2 cycles in the bridging FL cohort) of treatment and assessed by the investigator as not clearly related to the underlying disease: Any Grade 5 adverse event (AE; severity graded per NCI-CTCAE v4.0) unless due to the underlying malignancy or extraneous causes; AE of any grade that leads to a delay of more than (>)14 days in the start of the next treatment cycle; Grade 3 or 4 non-hematologic AEs (with exceptions); Lab results suggestive of potential drug-induced liver injury (according to Hy's law); Grade 3 or 4 neutropenia in the presence of sustained fever of >38 C (lasting >5 days) or a documented infection; Grade 4 neutropenia or thrombocytopenia lasting >7 days; Grade 3 or 4 thrombocytopenia if associated with Grade ≥3 bleeding; Other toxicities considered clinically relevant and related to study treatment as determined by the investigator and medical monitor.
Time Frame: Cycles 1, 2 (1 cycle is 28 days)
Population: Safety Population: participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Participants
  Any DLT | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
  Thrombocytopenia | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1

3. Secondary Outcome: Percentage of Participants With Complete Response at the End of Induction, Determined by the Investigator on the Basis of PET-CT Scans Using Modified Lugano 2014 Criteria
Description: The investigator evaluated responses at the end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT-based complete response (CR), which required a complete metabolic response with a score of 1, 2, or 3 with or without a residual mass in lymph nodes and extralymphatic sites on the PET 5-point scale for 18-fluorodeoxyglucose (FDG) uptake (1 = no uptake above background; 2 = uptake less than or equal to [≤] mediastinum; 3 = uptake greater than [>] mediastinum and ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly > liver and/or new lesions). The CR criteria were slightly modified to require normal bone marrow by morphology (if indeterminate, immunohistochemistry negative). PET-CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: ITT Population: all enrolled participants; exploratory analysis of the dose escalation phase (Phase 1). The study plan was for efficacy analyses to be based on responses in participants enrolled during the expansion phase (Phase 2), but it was not opened (i.e., no enrollment) and the study was terminated early.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Percentage of participants | 0 [0.00 to 77.64] | 33.3 [1.70 to 86.46] | 0 [0.00 to 77.64] | 0 [0.00 to 63.16] | 0 [0.00 to 52.71] | 50.0 [2.53 to 97.47] | 0 [0.00 to 52.71] | 40.0 [7.64 to 81.07]

4. Secondary Outcome: Percentage of Participants With Complete Response at the End of Induction, Determined by the Investigator on the Basis of PET-CT Scans Using Lugano 2014 Criteria
Description: The investigator evaluated responses at the end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT-based complete response (CR), which required a complete metabolic response with a score of 1, 2, or 3 with or without a residual mass in lymph nodes and extralymphatic sites on the PET 5-point scale for 18-fluorodeoxyglucose (FDG) uptake (1 = no uptake above background; 2 = uptake less than or equal to [≤] mediastinum; 3 = uptake greater than [>] mediastinum and ≤ liver; 4 = uptake moderately > liver; 5 = uptake markedly > liver and/or new lesions; X = new areas of uptake unlikely to be related to lymphoma). The CR criteria for participants with bone marrow involvement at screening required no evidence of FDG-avid disease in the marrow. PET-CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Percentage of participants | 0 [0.00 to 77.64] | 33.3 [1.70 to 86.46] | 0 [0.00 to 77.64] | 0 [0.00 to 63.16] | 0 [0.00 to 52.71] | 50.0 [2.53 to 97.47] | 0 [0.00 to 52.71] | 40.0 [7.64 to 81.07]

5. Secondary Outcome: Percentage of Participants With Complete Response at the End of Induction, Determined by the IRC on the Basis of CT Scans Alone Using Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a computed tomography (CT)-based complete response (CR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 centimetres in the longest transverse diameter of a lesion [LDi]; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 1
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Complete Response at the End of Induction, Determined by the Investigator on the Basis of CT Scans Alone Using Lugano 2014 Criteria
Description: The investigator evaluated responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a computed tomography (CT)-based complete response (CR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 centimetres in the longest transverse diameter of a lesion [LDi]; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). CT scans were performed at end of induction only on participants who had received at least 2 cycles of induction treatment; those without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Percentage of participants | 0 [0.00 to 77.64] | 33.3 [1.70 to 86.46] | 0 [0.00 to 77.64] | 0 [0.00 to 63.16] | 0 [0.00 to 52.71] | 0 [0.00 to 77.64] | 0 [0.00 to 52.71] | 20.0 [1.02 to 65.74]

7. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction, Determined by the IRC on the Basis of PET-CT Scans Using Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT-based objective response: either a complete (CR) or partial response (PR). A CR required a complete metabolic response with a score of 1, 2, or 3 on the PET 5-point scale (5PS) for 18-fluorodeoxyglucose (FDG) uptake (scores range from 1 [no uptake above background] to 5 [uptake markedly higher than liver and/or new lesions]), with or without a residual mass in lymph nodes and extralymphatic sites; and a PR required a partial metabolic response with a score of 4 or 5 on the 5PS with reduced 18-FDG uptake compared with baseline and residual mass(es) of any size. For bone marrow involvement, the CR criteria required no evidence of FDG-avid disease, and the PR criteria required residual uptake higher than in normal marrow but reduced compared with baseline. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 1
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction, Determined by the Investigator on the Basis of PET-CT Scans Using Lugano 2014 Criteria
Description: The investigator was to evaluate responses at the end of induction treatment using Lugano 2014 criteria for malignant lymphoma for a PET-CT-based objective response: either a complete (CR) or partial response (PR). A CR required a complete metabolic response with a score of 1, 2, or 3 on the PET 5-point scale (5PS) for 18-fluorodeoxyglucose (FDG) uptake (scores range from 1 [no uptake above background] to 5 [uptake markedly higher than liver and/or new lesions]), with or without a residual mass in lymph nodes and extralymphatic sites; and a PR required a partial metabolic response with a score of 4 or 5 on the 5PS with reduced 18-FDG uptake compared with baseline and residual mass(es) of any size. For bone marrow involvement, the CR criteria required no evidence of FDG-avid disease, and the PR criteria required residual uptake higher than in normal marrow but reduced compared with baseline. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: The study plan was for this efficacy analysis to be based on responses in participants enrolled during the expansion phase (Phase 2), but it was not opened (i.e., no enrollment) because the sponsor decided to terminate the study early due to the modest benefit achieved with the maximum tolerated dose during the dose escalation phase (Phase 1).
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction, Determined by an IRC on the Basis of CT Scans Alone Using Lugano 2014 Criteria
Description: The IRC was to evaluate responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a CT-based objective response: either a complete (CR) or partial response (PR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 cm in the LDi; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). The PR criteria required all of the following: a ≥50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites; no new lesions; non-measured lesion that is absent/normal, regressed, but no increase; and spleen must have regressed by >50% in length. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 1
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Objective Response at the End of Induction, Determined by the Investigator on the Basis of CT Scans Alone Using Lugano 2014 Criteria
Description: The investigator was to evaluate responses at the end of induction treatment using the Lugano 2014 response criteria for malignant lymphoma for a CT-based objective response: either a complete (CR) or partial response (PR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 cm in the LDi; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). The PR criteria required all of the following: a ≥50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites; no new lesions; non-measured lesion that is absent/normal, regressed, but no increase; and spleen must have regressed by >50% in length. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Within 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks; 1 cycle is 28 days)
Population: as for outcome 8
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Best Response of Complete Response or Partial Response During the Study, Determined by the Investigator on the Basis of CT Scans Alone Using Lugano 2014 Criteria
Description: The investigator was to evaluate responses throughout the study using the Lugano 2014 response criteria for malignant lymphoma for a CT-based best response of a complete (CR) or partial response (PR). The CR criteria required a complete radiologic response with all of the following: target nodes/nodal masses must regress to less than or equal to 1.5 cm in the LDi; no extralymphatic sites of disease; no non-measured or new lesions; enlarged organs regressing to normal size; and bone marrow normal by morphology (if indeterminate, immunohistochemistry negative). The PR criteria required all of the following: a ≥50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites; no new lesions; non-measured lesion that is absent/normal, regressed, but no increase; and spleen must have regressed by >50% in length. Participants without a post-baseline tumor assessment were to be considered non-responders.
Time Frame: Baseline, Cycle 2, end of induction (up to 6 cycles; 1 cycle is 28 days), every 2 months (FL) until end of maintenance or at 4 months (DLBCL) of consolidation treatment, and then every 6 months during follow-up until disease progression (up to 3.5 years)
Population: as for outcome 8
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Plasma Idasanutlin Concentrations in DLBCL and FL Participants at Nominal Sampling Timepoints Grouped by Idasanutlin Dose and Combination Partner (Obinutuzumab or Rituximab)
Description: The concentration of idasanutlin was determined using a validated assay. The duplication of the predose timepoint (0 hours) on Day 5 as an additional 24-hour timepoint on Day 5 was done in order to conduct pharmacokinetics analysis via non-compartmental analysis, and to derive idasanutlin exposure estimates up to the 24-hour post Day 5 dosing.
Time Frame: Predose (0 hours) and 6 hours postdose on Day 1 of Cycles 1, 2, and 4; Predose (0 hours) and 2, 4, 6, and 24 hours postdose on Day 5 of Cycles 1 and 2; Predose (0 hours) and 6 and 24 hours postdose on Cycle 4, Day 5 (1 cycle is 28 days)
Population: Pharmacokinetics Evaluable Population: all participants who received at least one dose of study drug. For this analysis, FL and DLBCL participants are grouped by idasanutlin dose and combination drug (obinutuzumab or rituximab). The number analyzed includes participants who were evaluable at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Groups:
- DLBCL/FL Combined: Idasanutlin 100 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) received induction treatment with idasanutlin 100 milligrams (mg) orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
- DLBCL/FL Combined: Idasanutlin 150 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) received induction treatment with idasanutlin 150 mg orally in combination with a fixed dose of obinutuzumab 1000 mg IV for 6 cycles (1 cycle = 28 days).
Arm/Group | DLBCL/FL Combined: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL/FL Combined: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 3 | 12 | 2 | 3 | 4
nanograms per millilitre (ng/mL)
  Cycle 1, Day 1: 0 hours: number analyzed (Participants) | 3 | 6 | 2 | 3 | 4
  Cycle 1, Day 1: 0 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1, Day 1: 6 hours: number analyzed (Participants) | 3 | 6 | 2 | 3 | 4
  Cycle 1, Day 1: 6 hours | 1540 (21.6) | 2210 (42.4) | 5540 (21.5) | 2130 (91.3) | 2980 (49.9)
  Cycle 1, Day 5: 0 hours: number analyzed (Participants) | 3 | 5 | 2 | 3 | 4
  Cycle 1, Day 5: 0 hours | 1150 (19.9) | 2150 (46.4) | 4120 (27.3) | 1660 (77.9) | 2920 (56.8)
  Cycle 1, Day 5: 2 hours: number analyzed (Participants) | 3 | 5 | 2 | 3 | 4
  Cycle 1, Day 5: 2 hours | 1230 (20.8) | 3570 (68.4) | 7850 (23) | 2970 (53.2) | 4970 (45.7)
  Cycle 1, Day 5: 4 hours: number analyzed (Participants) | 3 | 5 | 2 | 3 | 3
  Cycle 1, Day 5: 4 hours | 1670 (17.5) | 4360 (67.6) | 7930 (15.5) | 2910 (73.2) | 5910 (54.6)
  Cycle 1, Day 5: 6 hours: number analyzed (Participants) | 3 | 5 | 2 | 3 | 3
  Cycle 1, Day 5: 6 hours | 1730 (15.5) | 4220 (94.8) | 7310 (13.6) | 2820 (68.7) | 5200 (49.8)
  Cycle 1, Day 5: 24 hours: number analyzed (Participants) | 3 | 5 | 2 | 3 | 4
  Cycle 1, Day 5: 24 hours | 1150 (19.9) | 2150 (46.4) | 4120 (27.3) | 1660 (77.9) | 2920 (56.8)
  Cycle 2, Day 1: 0 hours: number analyzed (Participants) | 3 | 10 | 0 | 3 | 0
  Cycle 2, Day 1: 0 hours | 0 (0) | 0 (0) |  | 0 (0) |
  Cycle 2, Day 1: 6 hours: number analyzed (Participants) | 3 | 10 | 0 | 3 | 0
  Cycle 2, Day 1: 6 hours | 1660 (33.1) | 2480 (51.5) |  | 1260 (49.8) |
  Cycle 2, Day 5: 0 hours: number analyzed (Participants) | 0 | 7 | 0 | 2 | 0
  Cycle 2, Day 5: 0 hours |  | 2380 (27.2) |  | 2400 (67) |
  Cycle 2, Day 5: 2 hours: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  Cycle 2, Day 5: 2 hours |  | 4050 (54.9) |  |  |
  Cycle 2, Day 5: 4 hours: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0
  Cycle 2, Day 5: 4 hours |  | 4200 (38.2) |  |  |
  Cycle 2, Day 5: 6 hours: number analyzed (Participants) | 0 | 7 | 0 | 0 | 0
  Cycle 2, Day 5: 6 hours |  | 4010 (31.6) |  |  |
  Cycle 2, Day 5: 24 hours: number analyzed (Participants) | 0 | 7 | 0 | 0 | 0
  Cycle 2, Day 5: 24 hours |  | 2380 (27.2) |  |  |
  Cycle 4, Day 1: 0 hours: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Cycle 4, Day 1: 0 hours |  | 0 (0) |  |  |
  Cycle 4, Day 1: 6 hours: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Cycle 4, Day 1: 6 hours |  | 2730 (9.9) |  |  |
  Cycle 4, Day 5: 0 hours: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Cycle 4, Day 5: 0 hours |  | 2600 (25.6) |  |  |
  Cycle 4, Day 5: 6 hours: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Cycle 4, Day 5: 6 hours |  | 5210 (19.5) |  |  |
  Cycle 4, Day 5: 24 hours: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Cycle 4, Day 5: 24 hours |  | 2600 (25.6) |  |  |

13. Secondary Outcome: Serum Obinutuzumab Concentrations in DLBCL and FL Participants at Nominal Sampling Timepoints
Time Frame: Pre-infusion (0 hour) and 0.5 hours after end of obinutuzumab infusion on Day 1 of Cycles 1, 2, 4, and 6
Population: Pharmacokinetics Evaluable Population: all participants who received at least one dose of study drug. This analysis only includes FL and DLBCL participants who received obinutuzumab. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (μg/mL)
Groups:
- DLBCL/FL: Idasanutlin 100/150/200 mg + Obinutuzumab 1000 mg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma received induction treatment with idasanutlin 100 milligrams (mg), 150 mg, or 200 mg orally in combination with a fixed dose of obinutuzumab 1000 mg intravenously (IV) for 6 cycles (1 cycle = 28 days).
Arm/Group | DLBCL/FL: Idasanutlin 100/150/200 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 17
micrograms per millilitre (μg/mL)
  Cycle 1, Day 1: 0 hours: number analyzed (Participants) | 16
  Cycle 1, Day 1: 0 hours | 0 (0)
  Cycle 1, Day 1: 0.5 hours: number analyzed (Participants) | 13
  Cycle 1, Day 1: 0.5 hours | 397 (32.9)
  Cycle 2, Day 1: 0 hours: number analyzed (Participants) | 12
  Cycle 2, Day 1: 0 hours | 325 (59.8)
  Cycle 2, Day 1: 0.5 hours: number analyzed (Participants) | 12
  Cycle 2, Day 1: 0.5 hours | 703 (40.2)
  Cycle 4, Day 1: 0 hours: number analyzed (Participants) | 7
  Cycle 4, Day 1: 0 hours | 346 (46.1)
  Cycle 4, Day 1: 0.5 hours: number analyzed (Participants) | 7
  Cycle 4, Day 1: 0.5 hours | 685 (38.5)
  Cycle 6, Day 1: 0 hours: number analyzed (Participants) | 7
  Cycle 6, Day 1: 0 hours | 303 (49.5)
  Cycle 6, Day 1: 0.5 hours: number analyzed (Participants) | 7
  Cycle 6, Day 1: 0.5 hours | 639 (34.2)

14. Secondary Outcome: Serum Rituximab Concentrations in DLBCL Participants at Nominal Sampling Timepoints
Time Frame: Pre-infusion (0 hours) at Cycle 1, Day 1 and Cycle 2, Day 1; Post-infusion 0.5 hours at Cycle 1, Day 1 (1 cycle is 28 days)
Population: Pharmacokinetics Evaluable Population: all participants who received at least one dose of study drug. This analysis only includes DLBCL participants who received rituximab. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (μg/mL)
Groups:
- DLBCL Combined: Idasanutlin 150/200 mg + Rituximab 375 mg/m^2: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) received induction treatment with idasanutlin 150 mg or 200 mg orally in combination with rituximab 375 milligrams per square meter of body surface area (mg/m^2) IV for 6 cycles (1 cycle = 28 days).
Arm/Group | DLBCL Combined: Idasanutlin 150/200 mg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 7
micrograms per millilitre (μg/mL)
  Cycle 1, Day 1: 0 hours | 0 (0)
  Cycle 1, Day 1: 0.5 hours: number analyzed (Participants) | 6
  Cycle 1, Day 1: 0.5 hours | 197 (14.1)
  Cycle 2, Day 1: 0 hours: number analyzed (Participants) | 3
  Cycle 2, Day 1: 0 hours | 37.9 (58.1)

15. Secondary Outcome: Safety Summary of the Number of Participants With at Least One Adverse Event by Type and Severity According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0)
Description: The adverse event (AE) severity grading scale for the NCI CTCAE v4.0 was used for assessing AE severity. Any AEs that were not specifically listed in the NCI CTCAE, v4.0 were graded per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From first dose until 90 days after the last dose of study drug treatment (up to 31 months)
Population: Safety Population: participants who received at least one dose of any component of the combination treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Participants
  Any Adverse Event (AE) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
  Grade 5 AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3-5 AE | 1 | 3 | 2 | 2 | 3 | 1 | 3 | 4
  Serious AE | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 2
  AE Leading to any Study Treatment Discontinuation | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 2
  AE Leading to Dose Reductions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE Leading to Dose Interruptions | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1
  AE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related to Idasanutlin - Any AE | 1 | 2 | 2 | 2 | 4 | 1 | 4 | 5
  Related to Idasanutlin - Grade 3-5 AE | 1 | 2 | 2 | 1 | 2 | 1 | 3 | 4
  Related to Idasanutlin - Serious AE | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Related to Obinutuzumab - Any AE | 1 | 2 | 2 | 0 | 1 | 0 | 3 | 5
  Related to Obinutuzumab - Grade 3-5 AE | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 3
  Related to Obinutuzumab - Serious AE | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Related to Rituximab - Any AE | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Related to Rituximab - Grade 3-5 AE | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Related to Rituximab - Serious AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related AE Leading to Treatment Discontinuation | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1

16. Secondary Outcome: Baseline Value and Change From Baseline Values of Systolic Blood Pressure at Specified Timepoints
Description: Vital signs were measured prior to the infusion while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. Maint. = maintenance
Time Frame: Baseline, Days 1, 8, and 15 of Cycle 1, Day 1 of Cycles 2-6 (up to 6 cycles; 1 cycle is 28 days), and then every 2 months (FL) or every month (DLBCL) until end of maintenance or consolidation treatment, respectively (up to 29 months)
Population: Safety Population: participants who received at least one dose of any component of the combination treatment. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
millimeters of mercury (mmHg)
  Baseline (BL) - Value at Visit | 176.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 124.0 (7.9) | 107.5 (2.1) | 125.7 (39.4) | 119.0 (16.8) | 120.5 (17.7) | 109.3 (9.1) | 116.4 (10.5)
  Change from BL at Cycle 1 Day 1 | -34.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -2.0 (10.5) | -5.0 (4.2) | -2.7 (14.6) | -0.8 (10.6) | -3.5 (10.6) | 3.5 (9.4) | 4.8 (14.8)
  Change from BL at Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 5
  Change from BL at Cycle 1 Day 8 | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -5.0 (8.5) | -7.0 (8.5) |  |  | -6.5 (6.4) | -2.3 (15.2) | 6.4 (10.3)
  Change from BL at Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 2 | 3 | 5
  Change from BL at Cycle 1 Day 15 | 24.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -5.3 (14.6) |  |  |  | -3.5 (7.8) | 9.7 (13.4) | 8.0 (12.9)
  Change from BL at Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 5
  Change from BL at Cycle 2 Day 1 | -17.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -3.5 (19.1) |  | 0.0 (39.6) |  | -14.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 4.5 (4.9) | 8.6 (10.4)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 3
  Change from BL at Cycle 3 Day 1 | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 11.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  | -13.5 (3.5) | 10.5 (2.1) | 7.0 (8.9)
  Change from BL at Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Change from BL at Cycle 4 Day 1 | -22.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 12.5 (27.6) | 2.0 (1.4) | -10.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Change from BL at Cycle 5 Day 1 | -21.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 0.5 (4.9) | 12.5 (9.2) | 8.5 (9.2)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change from BL at Cycle 6 Day 1 |  |  |  |  |  | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 20.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.5 (0.7)
  Change from BL at Maint. Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 1 |  |  |  |  |  | -14.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 14.0 (9.9)
  Change from BL at Maint. Month 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 3 |  |  |  |  |  | 9.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 7.5 (10.6)
  Change from BL at Maint. Month 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 5 |  |  |  |  |  | -12.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 9.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 7 |  |  |  |  |  | -5.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 9 |  |  |  |  |  | -3.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 7.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 11 |  |  |  |  |  | -5.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 13 |  |  |  |  |  | -5.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 15 |  |  |  |  |  | -9.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 17 |  |  |  |  |  | -35.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 19 |  |  |  |  |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 21 |  |  |  |  |  | -21.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Follow-Up: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 2 | 4 | 4
  Change from BL at Follow-Up | -32.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -3.5 (9.2) | -25.0 (55.2) | -3.5 (0.7) | 9.5 (3.5) | 20.0 (15.5) | -1.3 (9.0)

17. Secondary Outcome: Baseline Value and Change From Baseline Values of Diastolic Blood Pressure at Specified Timepoints
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
millimeters of mercury (mmHg)
  Baseline (BL) - Value at Visit | 100.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 67.3 (12.1) | 72.0 (9.9) | 72.3 (12.3) | 70.3 (7.6) | 71.5 (9.2) | 76.3 (12.7) | 65.8 (6.9)
  Change from BL at Cycle 1 Day 1 | -17.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -2.0 (19.5) | -2.5 (2.1) | 7.3 (23.1) | -2.3 (7.4) | -2.0 (4.2) | 3.0 (4.9) | 6.4 (2.1)
  Change from BL at Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 5
  Change from BL at Cycle 1 Day 8 | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 1.3 (15.0) | -2.5 (6.4) |  |  | -2.0 (0.0) | -6.5 (1.3) | 9.2 (8.5)
  Change from BL at Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 2 | 3 | 5
  Change from BL at Cycle 1 Day 15 | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 3.0 (16.4) |  |  |  | 6.0 (4.2) | 0.0 (6.6) | 2.4 (8.3)
  Change from BL at Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 5
  Change from BL at Cycle 2 Day 1 | 7.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.0 (17.0) |  | 3.5 (13.4) |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -8.0 (2.8) | 12.0 (5.1)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 3
  Change from BL at Cycle 3 Day 1 | 3.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 3.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  | -5.5 (6.4) | -1.0 (4.2) | 5.3 (5.0)
  Change from BL at Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Change from BL at Cycle 4 Day 1 | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 3.0 (8.5) | -8.0 (7.1) | 7.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Change from BL at Cycle 5 Day 1 | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 3.5 (0.7) | -2.0 (7.1) | 2.5 (4.9)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change from BL at Cycle 6 Day 1 |  |  |  |  |  | 10.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 9.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 2.5 (3.5)
  Change from BL at Maint. Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 1 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 2.0 (0.0)
  Change from BL at Maint. Month 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 3 |  |  |  |  |  | 14.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 5.0 (8.5)
  Change from BL at Maint. Month 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 5 |  |  |  |  |  | -7.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -5.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 7 |  |  |  |  |  | 7.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 9 |  |  |  |  |  | 6.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 3.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 11 |  |  |  |  |  | -13.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 13 |  |  |  |  |  | 1.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 15 |  |  |  |  |  | 9.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 17 |  |  |  |  |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 19 |  |  |  |  |  | 7.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 21 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Follow-Up: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 2 | 4 | 4
  Change from BL at Follow-Up | -16.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -9.0 (21.2) | -15.5 (20.5) | 4.0 (4.2) | 10.5 (2.1) | 7.5 (20.2) | 9.3 (3.3)

18. Secondary Outcome: Baseline Value and Change From Baseline Values of Pulse Rate at Specified Timepoints
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
beats per minute
  Baseline (BL) - Value at Visit | 73.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 65.7 (1.2) | 100.5 (17.7) | 81.7 (3.1) | 76.0 (10.6) | 77.5 (12.0) | 79.5 (18.6) | 80.2 (9.9)
  Change from BL at Cycle 1 Day 1 | 10.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 15.7 (21.5) | -9.0 (8.5) | 0.0 (9.8) | 8.8 (12.0) | 2.5 (14.8) | 2.3 (6.4) | 9.0 (11.1)
  Change from BL at Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 5
  Change from BL at Cycle 1 Day 8 | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 11.0 (2.0) | -2.0 (1.4) |  |  | -0.5 (20.5) | 2.3 (6.4) | 9.0 (11.1)
  Change from BL at Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 2 | 3 | 5
  Change from BL at Cycle 1 Day 15 | -11.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 12.7 (13.4) |  |  |  | -3.5 (16.3) | -1.7 (13.1) | 3.2 (14.5)
  Change from BL at Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 5
  Change from BL at Cycle 2 Day 1 | 4.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 17.5 (17.7) |  | 7.0 (1.4) |  | -17.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -2.5 (4.9) | 6.4 (9.7)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 3
  Change from BL at Cycle 3 Day 1 | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 19.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  | -1.5 (16.3) | -4.5 (20.5) | -3.5 (10.6)
  Change from BL at Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Change from BL at Cycle 4 Day 1 | 1.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | -7.0 (12.7) | -5.0 (5.7) | 4.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Change from BL at Cycle 5 Day 1 | 15.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | -6.5 (10.6) | 3.0 (28.3) | 6.5 (4.9)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change from BL at Cycle 6 Day 1 |  |  |  |  |  | -1.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 31.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 15.0 (2.8)
  Change from BL at Maint. Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 1 |  |  |  |  |  | 6.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 10.0 (5.7)
  Change from BL at Maint. Month 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 3 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 2.0 (9.9)
  Change from BL at Maint. Month 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 5 |  |  |  |  |  | -5.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 11.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 7 |  |  |  |  |  | 1.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 9 |  |  |  |  |  | 6.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 11.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 11 |  |  |  |  |  | 18.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 13 |  |  |  |  |  | 11.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 15 |  |  |  |  |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 17 |  |  |  |  |  | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 19 |  |  |  |  |  | 1.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 21 |  |  |  |  |  | 13.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Follow-Up: number analyzed (Participants) | 1 | 0 | 2 | 2 | 2 | 2 | 4 | 4
  Change from BL at Follow-Up | 15.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -20.0 (18.4) | 11.5 (10.6) | 23.5 (20.5) | 15.0 (8.5) | 5.8 (14.8) | 10.3 (9.2)

19. Secondary Outcome: Baseline Value and Change From Baseline Values of Respiratory Rate at Specified Timepoints
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
breaths per minute
  Baseline (BL) - Value at Visit | 18.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 17.0 (2.6) | 19.0 (1.4) | 17.0 (1.7) | 17.0 (2.0) | 16.0 (0.0) | 16.0 (3.3) | 16.8 (3.0)
  Change from BL at Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 3
  Change from BL at Cycle 1 Day 1 | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.7 (1.2) | -1.0 (1.4) | -0.7 (1.2) | 0.3 (1.3) | 1.0 (1.4) | 2.3 (0.5) | 0.0 (0.0)
  Change from BL at Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 5
  Change from BL at Cycle 1 Day 8 | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -1.7 (2.1) | -1.0 (1.4) |  |  | 0.0 (0.0) | 2.0 (4.0) | 0.0 (2.4)
  Change from BL at Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 2 | 3 | 5
  Change from BL at Cycle 1 Day 15 | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -3.5 (2.1) |  |  |  | 1.0 (1.4) | 1.7 (1.5) | -0.2 (2.7)
  Change from BL at Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 4
  Change from BL at Cycle 2 Day 1 | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -2.5 (3.5) |  | 0.5 (0.7) |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 4.0 (5.7) | 0.0 (4.6)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 3
  Change from BL at Cycle 3 Day 1 | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  | 0.0 (0.0) | 4.0 (5.7) | -1.0 (4.2)
  Change from BL at Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Change from BL at Cycle 4 Day 1 | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 0.0 (0.0) | 2.0 (2.8) | 4.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Change from BL at Cycle 5 Day 1 | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 0.0 (0.0) | 1.0 (1.4) | 0.0 (5.7)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change from BL at Cycle 6 Day 1 |  |  |  |  |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 5.0 (NA) — Standard deviation could not be calculated from data for a single participant. | -2.0 (2.8)
  Change from BL at Maint. Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 1 |  |  |  |  |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -1.0 (4.2)
  Change from BL at Maint. Month 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 3 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -2.0 (2.8)
  Change from BL at Maint. Month 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 5 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 7 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 9 |  |  |  |  |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 11 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 13 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 15 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 17 |  |  |  |  |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 19 |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 21 |  |  |  |  |  | 2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Follow-Up: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 2 | 4 | 3
  Change from BL at Follow-Up | -2.0 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -2.0 (2.8) | -4.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.0 (2.8) | 1.0 (1.4) | 3.3 (3.2) | -0.7 (3.1)

20. Secondary Outcome: Baseline Value and Change From Baseline Values of Body Temperature at Specified Timepoints
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: degrees Celsius (C)
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
degrees Celsius (C)
  Baseline (BL) - Value at Visit | 36.60 (NA) — Standard deviation could not be calculated from data for a single participant. | 36.47 (0.45) | 36.35 (0.21) | 36.83 (0.15) | 36.58 (0.34) | 36.55 (0.21) | 36.50 (0.18) | 36.70 (3.3)
  Change from BL at Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 3
  Change from BL at Cycle 1 Day 1 | 0.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.00 (0.92) | -0.15 (0.21) | -0.07 (0.15) | 0.18 (0.33) | 0.05 (0.49) | 0.30 (0.22) | -0.18 (0.30)
  Change from BL at Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 5
  Change from BL at Cycle 1 Day 8 | 0.10 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.37 (0.50) | 0.95 (0.85) |  |  | 0.30 (0.28) | -0.13 (0.22) | 0.10 (0.45)
  Change from BL at Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 2 | 3 | 5
  Change from BL at Cycle 1 Day 15 | 0.10 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.20 (0.82) |  |  |  | 0.20 (0.28) | -0.23 (0.45) | -0.18 (0.26)
  Change from BL at Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 5
  Change from BL at Cycle 2 Day 1 | 0.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.10 (0.14) |  | -0.30 (0.14) |  | -0.50 (NA) — Standard deviation could not be calculated from data for a single participant. | -0.25 (0.49) | -0.04 (0.09)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 3
  Change from BL at Cycle 3 Day 1 | -0.20 (NA) — Standard deviation could not be calculated from data for a single participant. | -0.10 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  | -0.10 (0.42) | -0.50 (0.28) | -0.17 (0.21)
  Change from BL at Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Change from BL at Cycle 4 Day 1 | 0.00 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 0.05 (0.64) | 0.05 (0.21) | -0.10 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Change from BL at Cycle 5 Day 1 | 0.20 (NA) — Standard deviation could not be calculated from data for a single participant. |  |  |  |  | 0.35 (0.64) | -0.35 (0.49) | -0.20 (0.14)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change from BL at Cycle 6 Day 1 |  |  |  |  |  | 0.20 (NA) — Standard deviation could not be calculated from data for a single participant. | 0.20 (NA) — Standard deviation could not be calculated from data for a single participant. | -0.05 (0.21)
  Change from BL at Maint. Month 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 1 |  |  |  |  |  | 0.60 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -0.20 (0.14)
  Change from BL at Maint. Month 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Change from BL at Maint. Month 3 |  |  |  |  |  | 0.40 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -0.20 (0.57)
  Change from BL at Maint. Month 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 5 |  |  |  |  |  | 0.20 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -0.20 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 7 |  |  |  |  |  | 0.60 (NA) — Standard deviation could not be calculated from data for a single participant. |  | -0.10 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Change from BL at Maint. Month 9 |  |  |  |  |  | 0.30 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 0.20 (NA) — Standard deviation could not be calculated from data for a single participant.
  Change from BL at Maint. Month 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 11 |  |  |  |  |  | 0.70 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 13 |  |  |  |  |  | 0.40 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 15 |  |  |  |  |  | 0.70 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 17 |  |  |  |  |  | 0.40 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 19: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 19 |  |  |  |  |  | 0.80 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Maint. Month 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from BL at Maint. Month 21 |  |  |  |  |  | 0.50 (NA) — Standard deviation could not be calculated from data for a single participant. |  |
  Change from BL at Follow-Up: number analyzed (Participants) | 1 | 0 | 2 | 2 | 3 | 2 | 4 | 3
  Change from BL at Follow-Up | 0.10 (NA) — Standard deviation could not be calculated from data for a single participant. |  | 0.00 (0.14) | -0.40 (0.14) | 0.53 (0.71) | 0.30 (0.57) | -0.15 (0.47) | -0.10 (0.24)

21. Secondary Outcome: Number of Participants by Electrocardiogram (ECG) Results Assessment Shift From Baseline to Specified Post-Baseline Timepoints
Description: Single, resting, 12-lead ECG recordings were to be obtained after the participant had been resting in a supine position for at least 10 minutes. Any morphologic waveform changes or other ECG abnormalities were to be documented and clinical significance was determined based on the presence of symptoms, per the investigator's judgment. If the ECG assessment was missing at baseline then it was recorded as "Missing". The ECG results assessments are presented as the shift from baseline to post-baseline assessments at each timepoint. BL = baseline; Cyc1, D1 = Induction Cycle 1 Day 1; Cyc4, D1 = Induction Cycle 4 Day 1; CS = Clinically Significant; EOI = End of Induction Treatment - Completion/Discontinuation; EOM = End of Maintenance Treatment - Completion/Discontinuation; MM1 = Maintenance Month 1; Unsched = Unscheduled Visit
Time Frame: Baseline, Induction Cycle 1 Day 1 and Cycle 4 Day 1, End of Induction (up to 6 cycles; 1 cycle is 28 days); Every 2 months during maintenance treatment from Months 1-23; End of Maintenance (up to 24 months); Unscheduled Visits (as clinically indicated)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Participants
  Cyc1, D1: Normal (BL) to Normal: number analyzed (Participants) | 0 | 3 | 2 | 3 | 4 | 1 | 4 | 5
  Cyc1, D1: Normal (BL) to Normal |  | 1 | 1 | 0 | 2 | 0 | 4 | 2
  Cyc1, D1: Normal (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 3 | 2 | 3 | 4 | 1 | 4 | 5
  Cyc1, D1: Normal (BL) to Abnormal, not CS |  | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cyc1, D1: Abnormal, not CS (BL) to Normal: number analyzed (Participants) | 0 | 3 | 2 | 3 | 4 | 1 | 4 | 5
  Cyc1, D1: Abnormal, not CS (BL) to Normal |  | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Cyc1,D1: Abnormal, not CS (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 3 | 2 | 3 | 4 | 1 | 4 | 5
  Cyc1,D1: Abnormal, not CS (BL) to Abnormal, not CS |  | 1 | 1 | 1 | 2 | 1 | 0 | 2
  Cyc4, D1: Normal (BL) to Normal: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Cyc4, D1: Normal (BL) to Normal | 0 |  |  |  |  | 0 | 2 | 1
  Cyc4, D1: Normal (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Cyc4, D1: Normal (BL) to Abnormal, not CS | 1 |  |  |  |  | 0 | 0 | 0
  Cyc4, D1: Abnormal, not CS (BL) to Normal: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Cyc4, D1: Abnormal, not CS (BL) to Normal | 0 |  |  |  |  | 0 | 0 | 1
  Cyc4,D1: Abnormal, not CS (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Cyc4,D1: Abnormal, not CS (BL) to Abnormal, not CS | 0 |  |  |  |  | 1 | 0 | 0
  Cyc4, D1: Missing (BL) to Normal: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Cyc4, D1: Missing (BL) to Normal | 0 |  |  |  |  | 1 | 0 | 0
  EOI: Normal (BL) to Normal: number analyzed (Participants) | 1 | 2 | 2 | 1 | 3 | 2 | 3 | 3
  EOI: Normal (BL) to Normal | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 2
  EOI: Normal (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 2 | 2 | 1 | 3 | 2 | 3 | 3
  EOI: Normal (BL) to Abnormal, not CS | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOI: Abnormal, not CS (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 2 | 2 | 1 | 3 | 2 | 3 | 3
  EOI: Abnormal, not CS (BL) to Abnormal, not CS | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1
  EOI: Missing (BL) to Normal: number analyzed (Participants) | 1 | 2 | 2 | 1 | 3 | 2 | 3 | 3
  EOI: Missing (BL) to Normal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM1: Normal (BL) to Normal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  MM1: Normal (BL) to Normal |  |  |  |  |  |  |  | 1
  MM1: Abnormal, not CS (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  MM1: Abnormal, not CS (BL) to Abnormal, not CS |  |  |  |  |  |  |  | 1
  MM3: Abnormal, not CS (BL) to Normal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MM3: Abnormal, not CS (BL) to Normal |  |  |  |  |  |  |  | 1
  MM5: Abnormal, not CS (BL) to Normal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MM5: Abnormal, not CS (BL) to Normal |  |  |  |  |  |  |  | 1
  MM7: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM7: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM9: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM9: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM11: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM11: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM13: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM13: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM15: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM15: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM17: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM17: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM19: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM19: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM21: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM21: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  MM23: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MM23: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 |  |
  EOM: Normal (BL) to Normal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  EOM: Normal (BL) to Normal |  |  |  |  |  | 0 | 1 |
  EOM: Missing (BL) to Abnormal, not CS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  EOM: Missing (BL) to Abnormal, not CS |  |  |  |  |  | 1 | 0 |
  Unsched: Normal (BL) to Normal: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Unsched: Normal (BL) to Normal | 1 |  |  |  |  | 0 | 1 | 0
  Unsched: Normal (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Unsched: Normal (BL) to Abnormal, not CS | 0 |  |  |  |  | 0 | 1 | 0
  Unsched: Abnormal, not CS (BL) to Normal: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Unsched: Abnormal, not CS (BL) to Normal | 0 |  |  |  |  | 0 | 0 | 1
  Unsched: Abnormal, not CS (BL) to Abnormal, not CS: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Unsched: Abnormal, not CS (BL) to Abnormal, not CS | 0 |  |  |  |  | 1 | 0 | 0
  Unsched: Abnormal, not CS (BL) to Abnormal, CS: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Unsched: Abnormal, not CS (BL) to Abnormal, CS | 0 |  |  |  |  | 0 | 0 | 1

22. Secondary Outcome: Hematology Laboratory Test Results Shift Table: Number of Participants by Highest NCI-CTCAE v4.0 Grade at Baseline to Highest Grade Post-Baseline
Description: Clinical laboratory tests for hematology parameters were performed at local laboratories; any abnormal values (High or Low) were based on local laboratory normal ranges. Laboratory abnormalities are presented by the highest (worst) severity grade (according to NCI-CTCAE v4.0) at baseline to the highest grade post-baseline. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a medical intervention or a change in concomitant therapy. For a patient with multiple post-baseline abnormalities, the highest (worst) grade for a given lab test is reported. Abs. = absolute count; BL = baseline; WBC = white blood cell count
Time Frame: From Baseline until 35 days after the last dose of study drug (up to 29 months)
Population: Safety Population: participants who received at least one dose of any component of the combination treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Participants
  Hemoglobin (g/L), High: Grade (Gr.) 0 (BL) to 0 | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
  Hemoglobin (g/L), Low: Gr. 0 (BL) to 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hemoglobin (g/L), Low: Gr. 0 (BL) to 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  Hemoglobin (g/L), Low: Gr. 0 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hemoglobin (g/L), Low: Gr. 1 (BL) to 1 | 0 | 2 | 0 | 2 | 3 | 0 | 1 | 1
  Hemoglobin (g/L), Low: Gr. 1 (BL) to 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Hemoglobin (g/L), Low: Gr. 1 (BL) to 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/L), Low: Gr. 2 (BL) to 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hemoglobin (g/L), Low: Gr. 2 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin (g/L), Low: Gr. 3 (BL) to 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
  Lymphocytes Abs. (10^9/L), Low: Gr. 0 (BL) to 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Lymphocytes Abs. (10^9/L), Low: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 0 (BL) to 2 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 0 (BL) to 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 0 (BL) to 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 1 (BL) to 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes Abs. (10^9/L), Low: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 1 (BL) to 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 2 (BL) to 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 2 (BL) to 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes Abs. (10^9/L), Low: Gr. 3 (BL) to 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 3 (BL) to 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Lymphocytes Abs. (10^9/L), Low: Gr. 3 (BL) to 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Abs. (10^9/L), Low: Gr. 4 (BL) to 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophils,Total Abs (10^9/L),Low: Gr. 0(BL) to 0 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 2
  Neutrophils,Total Abs (10^9/L),Low: Gr. 0(BL) to 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neutrophils,Total Abs (10^9/L),Low: Gr. 0(BL) to 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Neutrophils,Total Abs (10^9/L),Low: Gr. 0(BL) to 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Neutrophils,Total Abs (10^9/L),Low: Gr. 0(BL) to 4 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1
  Neutrophils,Total Abs (10^9/L),Low: Gr. 2(BL) to 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets (10^9/L), Low: Gr. 0 (BL) to 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets (10^9/L), Low: Gr. 0 (BL) to 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
  Platelets (10^9/L), Low: Gr. 0 (BL) to 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets (10^9/L), Low: Gr. 0 (BL) to 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^9/L), Low: Gr. 0 (BL) to 4 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 1
  Platelets (10^9/L), Low: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets (10^9/L), Low: Gr. 1 (BL) to 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets (10^9/L), Low: Gr. 1 (BL) to 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBC (10^9/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
  WBC (10^9/L), Low: Gr. 0 (BL) to 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
  WBC (10^9/L), Low: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  WBC (10^9/L), Low: Gr. 0 (BL) to 2 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0
  WBC (10^9/L), Low: Gr. 0 (BL) to 3 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
  WBC (10^9/L), Low: Gr. 0 (BL) to 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  WBC (10^9/L), Low: Gr. 1 (BL) to 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (10^9/L), Low: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBC (10^9/L), Low: Gr. 1 (BL) to 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WBC (10^9/L), Low: Gr. 1 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

23. Secondary Outcome: Blood Chemistry Laboratory Test Results Shift Table: Number of Participants by Highest NCI-CTCAE v4.0 Grade at Baseline to Highest Grade Post-Baseline
Description: Clinical laboratory tests for blood chemistry parameters were performed at local laboratories; any abnormal values (High or Low) were based on local laboratory normal ranges. Laboratory abnormalities are presented by the highest (worst) severity grade (according to NCI-CTCAE v4.0) at baseline to the highest grade post-baseline. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a medical intervention or a change in concomitant therapy. For a patient with multiple post-baseline abnormalities, the highest (worst) grade for a given lab test is reported. BL = Baseline; Blood Gluc., Fast. = blood glucose, fasting; SGOT/AST = serum glutamic-oxaloacetic transaminase/aspartate transaminase; SGPT/ALT = serum glutamic-pyruvic transaminase/alanine transaminase; Triacylglyc. Lipase = triacylglycerol lipase
Time Frame: From Baseline until 35 days after the last dose of study drug (up to 29 months)
Population: Safety Population: participants who received at least one dose of any component of the combination treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 2 | 4 | 5
Participants
  Albumin (g/L), Low: Grade (Gr.) 0 (BL) to 0 | 1 | 3 | 2 | 1 | 2 | 2 | 4 | 3
  Albumin (g/L), Low: Grade (Gr.) 0 (BL) to 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Albumin (g/L), Low: Grade (Gr.) 0 (BL) to 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Albumin (g/L), Low: Grade (Gr.) 1 (BL) to 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Alkaline Phosphatase (U/L), High: Gr. 0 (BL) to 0 | 0 | 3 | 2 | 2 | 3 | 1 | 4 | 3
  Alkaline Phosphatase (U/L), High: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Alkaline Phosphatase (U/L), High: Gr. 1 (BL) to 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Amylase (U/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 1 | 2 | 3 | 5
  Amylase (U/L), High: Missing (BL) to Gr. 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Amylase (U/L), High: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin (umol/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 4 | 2 | 3 | 5
  Bilirubin (umol/L), High: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Blood Gluc,Fast(mmol/L), High: Missing(BL) to Gr 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Blood Gluc,Fast(mmol/L), High: Gr. 0(BL) to 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Gluc,Fast(mmol/L), High: Gr. 1 (BL) to 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Gluc,Fast(mmol/L), High: Missing(BL) to Gr 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Gluc.,Fast.(mmol/L), High: Missing (All) | 0 | 3 | 0 | 3 | 4 | 1 | 3 | 4
  Blood Gluc,Fast(mmol/L), Low: Gr. 0 (BL) to 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Blood Gluc,Fast(mmol/L), Low: Missing(BL) to Gr 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Blood Gluc.,Fast.(mmol/L), Low: Missing (All) | 0 | 3 | 0 | 3 | 4 | 1 | 3 | 4
  Calcium (mmol/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 3 | 2 | 4 | 5
  Calcium (mmol/L), High: Gr. 1 (BL) to 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium (mmol/L), Low: Gr. 0 (BL) to 0 | 1 | 2 | 2 | 2 | 3 | 2 | 3 | 4
  Calcium (mmol/L), Low: Gr. 0 (BL) to 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Calcium (mmol/L), Low: Gr. 0 (BL) to 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Calcium (mmol/L), Low: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine (umol/L), High: Gr. 0 (BL) to 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 3
  Creatinine (umol/L), High: Gr. 0 (BL) to 1 | 0 | 1 | 2 | 2 | 2 | 2 | 1 | 1
  Creatinine (umol/L), High: Gr. 0 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine (umol/L), High: Gr. 1 (BL) to 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine (umol/L), High: Gr. 1 (BL) to 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine (umol/L), High: Gr. 1 (BL) to 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Glucose (mmol/L), High: Gr. 0 (BL) to 0 | 0 | 3 | 0 | 3 | 4 | 2 | 4 | 5
  Glucose (mmol/L), High: Missing (BL) to Gr. 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose (mmol/L), High: Gr. 0 (BL) to 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mmol/L), High: Missing (All) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose (mmol/L), Low: Gr. 0 (BL) to 0 | 1 | 2 | 0 | 2 | 4 | 2 | 4 | 4
  Glucose (mmol/L), Low: Missing (BL) to Gr. 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose (mmol/L), Low: Gr. 0 (BL) to 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Glucose (mmol/L), Low: Missing (All) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Phosphorus (mmol/L), Low: Gr. 0 (BL) to 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 2
  Phosphorus (mmol/L), Low: Missing (BL) to Gr. 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1
  Phosphorus (mmol/L), Low: Missing (BL) to Gr. 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Phosphorus (mmol/L), Low: Missing (All) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2
  Potassium (mmol/L), High: Gr. 0 (BL) to 0 | 0 | 3 | 2 | 2 | 4 | 2 | 4 | 5
  Potassium (mmol/L), High: Gr. 0 (BL) to 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium (mmol/L), Low: Gr. 0 (BL) to 0 | 1 | 2 | 2 | 3 | 3 | 2 | 4 | 3
  Potassium (mmol/L), Low: Gr. 0 (BL) to 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium (mmol/L), Low: Gr. 2 (BL) to 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (mmol/L), Low: Gr. 2 (BL) to 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  SGOT/AST (U/L), High: Gr. 0 (BL) to 0 | 1 | 2 | 2 | 2 | 4 | 2 | 4 | 5
  SGOT/AST (U/L), High: Gr. 1 (BL) to 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  SGPT/ALT (U/L), High: Gr. 0 (BL) to 0 | 1 | 2 | 1 | 3 | 2 | 2 | 4 | 5
  SGPT/ALT (U/L), High: Gr. 1 (BL) to 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  SGPT/ALT (U/L), High: Gr. 1 (BL) to 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Sodium (mmol/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 3 | 2 | 4 | 4
  Sodium (mmol/L), High: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium (mmol/L), High: Gr. 1 (BL) to 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Sodium (mmol/L), Low: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 2 | 4 | 2 | 4 | 3
  Sodium (mmol/L), Low: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Sodium (mmol/L), Low: Gr. 0 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium (mmol/L), Low: Gr. 1 (BL) to 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Triacylglyc. Lipase (U/L), High: Gr. 0 (BL) to 0 | 0 | 3 | 2 | 3 | 2 | 1 | 3 | 4
  Triacylglyc. Lipase (U/L), High: Gr. 0 (BL) to 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Triacylglyc. Lipase (U/L), High: Gr. 0 (BL) to 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triacylglyc Lipase (U/L),High: Missing(BL) to Gr 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Triacylglyc Lipase (U/L),High: Missing(BL) to Gr 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Uric Acid (umol/L), High: Gr. 0 (BL) to 0 | 1 | 3 | 2 | 3 | 2 | 2 | 3 | 4
  Uric Acid (umol/L), High: Missing(BL) to Gr. 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Uric Acid (umol/L), High: Gr. 0 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Uric Acid (umol/L), High: Gr. 3 (BL) to 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Uric Acid (umol/L), High: Gr. 4 (BL) to 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose until 90 days after the last dose of study drug treatment (up to 31 months), except for serious AEs related to treatment
Description: Investigators seek information on adverse events (AEs) at each patient contact. All AEs were recorded, regardless of who reported them. After informed consent but prior to initiation of study drug, only serious AEs caused by protocol-mandated intervention were to be reported. After initiation of study drug, all AEs were to be reported until 90 days after the last dose of study drug. After this period, only serious AEs believed to be related to prior study drug treatment were to be reported.
Arm/Group | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/3 | 2/2 | 2/3 | 2/4 | 0/2 | 0/4 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 1/2 | 0/3 | 2/4 | 1/2 | 1/4 | 2/5
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2 | 3/3 | 4/4 | 2/2 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (N=1) | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=3) | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg (N=2) | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 (N=3) | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 (N=4) | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (N=2) | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=4) | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLBCL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (N=1) | DLBCL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=3) | DLBCL Non-Bridging: Idasanutlin 200 mg + Obinutuzumab 1000 mg (N=2) | DLBCL Bridging: Idasanutlin 150 mg + Rituximab 375 mg/m^2 (N=3) | DLBCL Bridging: Idasanutlin 200 mg + Rituximab 375 mg/m^2 (N=4) | FL Non-Bridging: Idasanutlin 100 mg + Obinutuzumab 1000 mg (N=2) | FL Non-Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=4) | FL Bridging: Idasanutlin 150 mg + Obinutuzumab 1000 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 4 (4) | 1 (2) | 3 (10) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 4 (7) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 1 (4) | 3 (8) | 3 (5)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (6) | 3 (8) | 5 (11)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (8) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophilus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the overall modest benefit achieved with the maximum tolerated dose during the dose escalation phase, the Sponsor decided not to open the expansion phase and terminated the study. Consequently, some planned analyses could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT02624986/Prot_SAP_000.pdf